CLINICAL TRIAL: NCT02420223
Title: Randomized Controlled Pilot Study Using Propranolol to Decrease Gene Expression of Stress-Mediated Beta-Adrenergic Pathways in Hematopoietic Stem Cell Transplant (HCT) Recipients
Brief Title: Study of Propranolol to Decrease Gene Expression of Stress-Mediated Beta-Adrenergic Pathways in HCT Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jennifer M. Knight, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00024391
Record Dates: First submitted 2015-03-03; First posted 2015-04-17 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: Recipients
MeSH Terms: conditions — Multiple Myeloma | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Patient's randomized to the Propranolol arm will be starting 7 days prior to transplant and continuing through 28 days post-transplant. Propranolol will start at 20mg twice daily and will be titrated to 40mg twice daily as tolerated. Both groups will come back to the hospital weekly in order to assess items such as patient's level of anxiety, depression, your adherence, and also to monitor for side effects. The patient's will complete questionnaires during your visit. These will take approximately 15 minutes to complete. This will continue for up to 7 total weeks for patient's on the Propranolol arm.
  Interventions: Drug: Propranolol
- Control Arm (No Intervention): Both groups will come back to the hospital weekly in order to assess items such as patient's level of anxiety, depression, your adherence, and also to monitor for side effects. The patient's will complete questionnaires during your visit. These will take approximately 15 minutes to complete. This will continue for 6 total weeks for patient's on the control arm.

INTERVENTIONS:
Drug: Propranolol
  Other Names: Hemangeol, Inderal LA, Inderal XL, InnoPran XL, Inderal
  Arms: Propranolol

SUMMARY:
This is a randomized controlled pilot study designed to evaluate whether the beta-adrenergic antagonist propranolol is effective in decreasing gene expression of stress-mediated beta-adrenergic pathways among a cohort of individuals receiving an autologous hematopoietic stem cell transplant (HCT) for multiple myeloma.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study designed to evaluate whether a drug designed to block the physiologic effects of stress is effective at blocking stress-related gene expression in people receiving autologous stem cell transplants (their own cells) for multiple myeloma. Such stress-related gene expression is one way that the body is programmed to make specific proteins under conditions of stress. These proteins are believed to contribute to worse health outcomes. By using the drug propranolol, we aim to see whether we might block these negative health effects of stress as occur in the cancer setting and during the transplant process. We hypothesize that individuals taking propranolol will have more favorable gene expression.

We will enroll 40 individuals, randomizing half to receive propranolol and half to serve as the control group not on the study drug. Study participants will start propranolol three weeks prior to their transplant and continue it until 30 days after the transplant. We will explore the effect of socioeconomic status, depression, and anxiety on individuals' gene expression response to propranolol with the idea that the more impoverished, anxious, or depressed individuals will display an even greater change in their gene expression. Part of the purpose of this study is also be to assess whether it is feasible to give this drug to individuals with cancer. Results of this study may inform larger trials assessing the effects of propranolol on cancer progression.

ELIGIBILITY:
Inclusion Criteria:

Patients with multiple myeloma receiving an autologous HCT are eligible when the following criteria are met:

1. 18-75 years of age
2. ≤ 1 year since initiation of systemic anti-myeloma therapy
3. Patient is scheduled for autologous hematopoietic stem cell transplant as the upfront therapy for their multiple myeloma
4. Karnofsky Performance Status of ≥90 %; patients eligible for HCT are eligible for the study
5. All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile.

Exclusion Criteria:

1. Prior autologous HCT
2. Non secretory multiple myeloma
3. Concurrent beta-blocker therapy at or within 3 weeks of study entry.
4. Previous intolerance to beta-blocker therapy
5. Any medical contraindications to beta-blocker therapy including, but not limited to, symptomatic hypotension; drug hypersensitivity; sinus bradycardia, sick sinus syndrome, or 2nd or 3rd degree atrioventricular block without a pacemaker; uncompensated heart failure; or uncontrolled asthma
6. Active, untreated depression screened for by the HCT physician (Patients who screen positive will be offered a referral to the Medical College of Wisconsin Psycho-Oncology program for further evaluation and treatment)
7. Concurrent use of medications as specified in the protocol throughout the study or within one week of study entry.
8. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knight, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knight JM, Rizzo JD, Hari P, Pasquini MC, Giles KE, D'Souza A, Logan BR, Hamadani M, Chhabra S, Dhakal B, Shah N, Sriram D, Horowitz MM, Cole SW. Propranolol inhibits molecular risk markers in HCT recipients: a phase 2 randomized controlled biomarker trial. Blood Adv. 2020 Feb 11;4(3):467-476. doi: 10.1182/bloodadvances.2019000765. PMID 32027744
- [Derived] Knight JM, Kerswill SA, Hari P, Cole SW, Logan BR, D'Souza A, Shah NN, Horowitz MM, Stolley MR, Sloan EK, Giles KE, Costanzo ES, Hamadani M, Chhabra S, Dhakal B, Rizzo JD. Repurposing existing medications as cancer therapy: design and feasibility of a randomized pilot investigating propranolol administration in patients receiving hematopoietic cell transplantation. BMC Cancer. 2018 May 24;18(1):593. doi: 10.1186/s12885-018-4509-0. PMID 29793446

RESULTS

PARTICIPANT FLOW:
Groups:
- Propranolol: Patient's randomized to the Propranolol arm will be starting 7 days prior to transplant and continuing through 28 days post-transplant. Propranolol will start at 20mg twice daily and will be titrated to 40mg twice daily as tolerated. Both groups will come back to the hospital weekly in order to assess items such as patient's level of anxiety, depression, your adherence, and also to monitor for side effects. The patient's will complete questionnaires during your visit. These will take approximately 15 minutes to complete. This will continue for up to 7 total weeks for patient's on the Propranolol arm.
  Propranolol
Period: Overall Study
Arm/Group | Propranolol | Control Arm
Started | 12 | 13
Completed | 11 | 11
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Control Arm | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.1) | 63 (8.6) | 61 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Beta-adrenergically Mediated Gene Expression (Change From Baseline)
Description: Expression (up or down regulation) of genes involved in the stress response can be modulated through the beta-adrenergic pathway. The log2 RNA abundance is a means to normalize results to determine whether a gene is up regulated (value greater than 1) or down regulated (value less than 1). Differential change in log2 RNA abundance is defined by the fold change (FC) as log2FC=Log2(B)-Log2(A). Logarithmic measures are unitless. The change in the measure between two time points determines whether a gene has up-or down-regulated.
Time Frame: Baseline (Pre-Transplant); 4 weeks post-transplant
Measure: Mean (Standard Error); unit: Unitless
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Unitless | -0.407 (0.165) | 0.0099 (0.103)
Statistical Analysis 1: Comparison: Propranolol; Test type: Superiority; p = .017, Regression, Logistic
Statistical Analysis 2: Comparison: Control Arm; Test type: Superiority; p = 0.337, Regression, Logistic

2. Secondary Outcome: Patient-reported Depression and Anxiety Scores
Description: This measure will be assessed using the Hospital Anxiety and Depression Scale (HADS). The HADS scale includes fourteen 4-response Likert-scale questions graded 0 to 3. Seven questions are specific to depression; 7 questions are specific to anxiety. The score is the total of the responses in their respective categories. Lower scores indicated less depression and/or anxiety. Scores 0-7 indicate normal status; scores 8-10 suggest borderline abnormal status; and scores 11-21 indicate abnormal status. Only anxiety scores are presented.
Time Frame: Baseline and 4 weeks
Population: One propranolol subject was discontinued due to symptomatic hypotension. Two control subjects were discontinued doe to initiation of beta-blocker therapy for cardiac arrhythmia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline Anxiety Score | 7.3 (3.5) | 7.4 (3.7)
  4-Week Anxiety Score: number analyzed (Participants) | 11 | 11
  4-Week Anxiety Score | 4.4 (2.3) | 5.2 (3.7)

3. Secondary Outcome: Number of Subjects Experiencing Engraftment Syndrome as a Function of Beta-blocker Administration
Description: Number of subjects experiencing any of: fever, diarrhea or rash requiring steroid intervention within 48 hours before or after neutrophil recovery.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Participants | 6 | 3

4. Secondary Outcome: Time (Days) to Neutrophil Engraftment
Description: This measure is the mean time to the beginning of three consecutive days where the neutrophil count (absolute neutrophil count) was 500 cells/mm^3 (0.5 x 10^9/L) or greater.
Time Frame: 4 weeks after transplant
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Days | 10.5 (1.0) | 11.9 (3.7)
Statistical Analysis 1: Comparison: Propranolol vs Control Arm; Test type: Superiority; p = 0.14, t-test, 2 sided

5. Secondary Outcome: Time (Days) to Platelet Engraftment
Description: This measure is the mean time to the beginning of three consecutive days where the platelet count is at least 20,000/mm^3 (20 x 10^9/L) unsupported by a platelet transfusion.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Days | 16.6 (4.1) | 19.6 (5.4)
Statistical Analysis 1: Comparison: Propranolol vs Control Arm; Test type: Superiority; p = 0.41, t-test, 2 sided

6. Secondary Outcome: Number of Participants Diagnosed With Culture-positive Infection or Neutropenic Fever Greater Than 100.4 Degrees Fahrenheit
Description: This measure is the number of subjects diagnosed with culture-positive infection or neutropenic fever greater than 100.4 degrees Fahrenheit.
Time Frame: Up to 100 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Participants | 1 | 6
Statistical Analysis 1: Comparison: Propranolol vs Control Arm; Test type: Superiority; p = 0.06, Likelihood ration Chi-Square test

7. Secondary Outcome: Number of Participants With Myeloma Response as a Function of Beta-blocker Administration
Description: This measure is the number of participants experiencing a response defined by the International Uniform Response Criteria as: very good partial response (VGPR) or better (near complete response (nCR), complete response (CR), and stringent CR (sCR) according to at day 100 post-Hematopoietic Cell Transplant.
Time Frame: 100 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Control Arm
Number analyzed (Participants) | 12 | 13
Participants
  Stable Disease | 1 | 0
  Partial Response | 5 | 5
  Very Good Partial Response | 5 | 5
  Complete Response | 1 | 3

ADVERSE EVENTS:
Time Frame: 100 Days
Arm/Group | Propranolol | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/13
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=12) | Control Arm (N=13)
Edema of limb (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=12) | Control Arm (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT02420223/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT02420223/ICF_001.pdf